CLINICAL TRIAL: NCT04860791
Title: Validation Study of the French Adaptation of the MSWDQ-23 Questionnaire, a Tool Assessing the Work Difficulties of Patients With Multiple Sclerosis.
Brief Title: Validation of the French Adaptation of the MSWDQ-23 Questionnaire
Acronym: WORKSEP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20-PP-03
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Sclerosis patients
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Patients will complete the MSWDQ-23 in French, as well as the DEX, questionnaire for the evaluation of executive dysfunction in daily life, to evaluate their cognitive complaints and the SF36 questionnaire to evaluate their quality of life

SUMMARY:
MS is an autoimmune disease of the central nervous system that affects more than 120,000 people in France. The average age of onset of the disease is between 25 and 35 years. Given the wide range of ages of the patients, from 4 to 80 years, the ethical and socio-economic stakes are high in order to maintain their autonomy, sociability, family and intimate life, and their employment in the best possible conditions and for as long as possible.

However, to date, there are no evaluation tools in French that allow us to understand the difficulties at work of MS patients.

The Multiple Sclerosis Work Difficulties Questionnaire (MSWDQ-23) was developed specifically for MS patients and validated in English [1]. There is a short version of this questionnaire that facilitates its use in clinical practice [2]. It has been translated and validated in Spanish through a multicenter study, and is currently being validated in German, but does not currently exist in French [3]. The main objective of the WORKSEP project is to validate the French version of this questionnaire through a multicenter population-based cohort within the framework of the French-speaking Multiple Sclerosis Society (SFSEP). This validation study will involve the inclusion of 206 French-speaking MS patients, regardless of their professional status, all forms of MS combined, from the early stage (Clinically Isolated Syndrome) to the more advanced stages (primary and secondary progressive forms).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old.
* Native French speaker.
* A diagnosis of Clinically Isolated Syndrome or MS defined according to the 2017 McDonald criteria.
* Be affiliated with the social security system.
* Agree to participate in the study.

Exclusion Criteria:

Opposition to the use of the data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French-speaking MS patients with or without cognitive complaints and regardless of their occupational status will be prospectively recruited at their scheduled disease follow-up consultation
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
MSWDQ-23 score | 1 day
  total score out of 100

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Besancon University Hospital, Besançon
  - Bordeaux university hospital, Bordeaux
  - Caen university hospital, Caen
  - Clermont Ferrand university hospital, Clermont-Ferrand
  - Gonesse hospital, Gonesse
  - Libourne hospital, Libourne
  - Lille University Hospital, Lille
  - Groupement des Hôpitaux de l'Institut Catholique de Lille, Lomme
  - Lyon University Hospital, Lyon
  - Marseille University Hospital, Marseille
  - Nancy Hospital, Nancy
  - Nimes university hospital, Nîmes
  - APHP, Paris
  - Rouen univestity hospital, Rouen
  - Saint Etienne University Hospital, Saint-Etienne
  - Strasnourg university hospital, Strasbourg

IPD SHARING:
Plan to Share IPD: No